CLINICAL TRIAL: NCT04285216
Title: Combined Effects of Dry Needling and Strain Counter Strain Technique in Myofascial Trigger Points of Upper Trapezius
Brief Title: Effects of Dry Needling and Strain Counter Strain Technique in Myofascial Trigger Points of Upper Trapezius
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MSOMPT/Spring19/031 Aqsa Aroob
Record Dates: First submitted 2020-02-11; First posted 2020-02-26 (Actual); Last update posted 2020-09-22 (Actual); Status verified 2020-09

CONDITIONS: Trigger Point Pain, Myofascial
Keywords: Dry needling; Myofascial trigger points; Upper Trapezius; Strain counter strain
MeSH Terms: conditions — Myofascial Pain Syndromes | interventions — Dry Needling

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Outcome Assessor will be binded
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dry needling (Experimental): Hot pack 10 mints,stretching,Neck isometrics, dry needling(DN) and Strain counterstrain(SCS)
  Interventions: Other: Dry Needling
- Strain counter strain (Active Comparator): Hot pack 10 minutes, stretching,Neck isometrics, Strain counter strain (S C S)
  Interventions: Other: Strain counter strain

INTERVENTIONS:
Other: Dry Needling — Hot pack 10 mints,stretching,Neck isometrics, dry needling(DN) and Strain counterstrain(SCS)
  Arms: Dry needling
Other: Strain counter strain — Hot pack 10 mints, stretchings,Neck isometrics, Strain counterstrain(SCS)
  Arms: Strain counter strain

SUMMARY:
To determine the effects of Dry Needling and Strain Counter Strain Technique in Myofascial Trigger Points of Upper Trapezius

DETAILED DESCRIPTION:
It is Randomized Controlled trail will be conduct in Mayo Hospital Lahore and Alnoor Hospital Awan town Lahore. Non probability consecutive sampling technique will be used to collect the data. Each group contain the 14 patients, Patient will be divided into two groups. Group A will be experimental group treated by Dry needling and strain counter strain with baseline treatment and Group B will be control group treated by Strain counter strain with baseline treatment(Hot pack 10 mints,stretching,Neck isometrics). Neck Disability index (NDI) ,visual analogue scale(VAS) and goniometer will be used as data collecting tools.

ELIGIBILITY:
Inclusion Criteria:

* Patients with non-specific neck pain, having active myofascial trigger points in upper trapezius muscle.
* Patient of both gender under the age of 20-40 year
* bilateral pain involving the upper trapezius
* a duration of pain of at least 3 months
* pain localized in the cervical and occipital regions but not in the orofacial region.
* restricted cervical range of motion(side flexion)

Exclusion Criteria:

* history of traumatic injuries (e.g., contusion, fracture, and whiplash injury)
* needle phobia patients.
* systemic diseases such as blood coagula tion disorders, chronic pain syndrome, cancer,allergies fibromyalgia, systemic lupus erythematous, and psoriatic arthritis.
* cervical spine surgery patients.
* orofacial pain and temporomandibular disorders
* neurologic disorders (e.g., trigeminal neuralgia or occipital neuralgia)
* medical diagnosis of any primary headache (tension type or migraine) clinical diagnosis of cervical radiculopathy or myelopathy
* history of previous physical therapy intervention for the cervical region in last 6 month
* use of anticoagulants, opioids or antiepileptic medications

Ages: 20 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 28 (Actual)
Dates: Start 2019-09-15 (Actual); Primary Completion 2020-06-20 (Actual); Study Completion 2020-08-28 (Actual)

PRIMARY OUTCOMES:
Numeric Pain Rating Scale (NPRS) | 4 months
  The Numerical Pain Rating Scale (NPRS) is a subjective measure in which individuals rate their pain on an eleven-point numerical scale. The scale is composed of 0 (no pain at all) to 10 (worst imaginable pain).
Range of Motion | 4 months
  Standard Goniometer will be used.Higher score shows improvement.

SECONDARY OUTCOMES:
Disability | 4 months
  Scoring: For each section the total possible score is 5: if the first statement is marked the section score = 0, if the last statement is marked it = 5. If all ten sections are completed the score is calculated as follows: Example:16 (total scored) 50 (total possible score) x 100 = 32% If one section is missed or not applicable the score is calculated: 16 (total scored) 45 (total possible score) x 100 = 35.5% Minimum Detectable Change (90% confidence): 5 points or 10 %points

CONTACTS AND LOCATIONS:
Overall Officials: Maryam Shabbir, Phd, Principal Investigator — Riphah International University
Locations (1):
- Mayo Hospital, Lahore, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gerwin RD, Shannon S, Hong CZ, Hubbard D, Gevirtz R. Interrater reliability in myofascial trigger point examination. Pain. 1997 Jan;69(1-2):65-73. doi: 10.1016/s0304-3959(96)03248-4. PMID 9060014
- [Background] Lavelle ED, Lavelle W, Smith HS. Myofascial trigger points. Anesthesiol Clin. 2007 Dec;25(4):841-51, vii-iii. doi: 10.1016/j.anclin.2007.07.003. PMID 18054148
- [Background] Fischer AA. Pressure algometry over normal muscles. Standard values, validity and reproducibility of pressure threshold. Pain. 1987 Jul;30(1):115-126. doi: 10.1016/0304-3959(87)90089-3. PMID 3614975
- [Background] Kalichman L, Vulfsons S. Dry needling in the management of musculoskeletal pain. J Am Board Fam Med. 2010 Sep-Oct;23(5):640-6. doi: 10.3122/jabfm.2010.05.090296. PMID 20823359
- [Background] Tough EA, White AR, Cummings TM, Richards SH, Campbell JL. Acupuncture and dry needling in the management of myofascial trigger point pain: a systematic review and meta-analysis of randomised controlled trials. Eur J Pain. 2009 Jan;13(1):3-10. doi: 10.1016/j.ejpain.2008.02.006. Epub 2008 Apr 18. PMID 18395479
- [Background] avaid HMW, Ahmad A, Ajmad F, Liaqat S, Tahir S. Effects of conventional physical therapy with or without strain counterstrain in patients with trigger points of upper trapezius; a randomized controlled clinical trial. Annals of King Edward Medical University. 2016;22(3).
- [Background] Somprasong S, Mekhora K, Vachalathiti R, Pichaiyongwongdee S. Effects of strain counter-strain and stretching techniques in active myofascial pain syndrome. Journal of physical therapy science. 2011;23(6):889-93.